CLINICAL TRIAL: NCT02284789
Title: Content and Psychometric Validation Study of the Colorado Adult Joint Assessment Scale (CAJAS) in Subjects With Moderate to Severe Hemophilia A Treated on Prophylaxis
Brief Title: Colorado Adult Joint Assessment Scale (CAJAS) Validation
Acronym: CAJAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 17819
Record Dates: First submitted 2014-11-04; First posted 2014-11-06 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Hemophilia A
Keywords: Hemophilia
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CAJAS evaluation (Other)
  Interventions: Other: Colorado Adult Joint Assessment Evaluation

INTERVENTIONS:
Other: Colorado Adult Joint Assessment Evaluation — Physical evaluation of 6 joints, ankles, knees and elbows

SUMMARY:
To obtain evidence of content validity and reliability of the Colorado Adult Joint Assessment Scale (CAJAS), a clinician-reported outcome (ClinRO) measure, as adapted for use in a population of adults with moderate to severe hemophilia A treated with coagulation factor VIII (FVIII) therapy as secondary prophylaxis or episodic treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male, 18 to 50 years of age
* Diagnosis of moderate to severe hemophilia A (documented <1-2% Factor VIII Concentration [FVIII:C])
* Willing to maintain current FVIII treatment regimen, whether prophylactic or on-demand, for the duration of the study

Exclusion Criteria:

* Routine need for wheelchair or routine need for two canes or crutches
* Diagnosis of another bleeding disorder such as von Willebrand Disease
* Known event that would interfere with the scheduled CAJAS evaluations (e.g., elective joint surgery, vacation)

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2015-02; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Colorado Adult Joint Assessment Score (CAJAS) | Up to 25 days

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (4):
- United States (4):
  - Orange, California
  - Aurora, Colorado
  - Indianapolis, Indiana
  - Portland, Oregon